CLINICAL TRIAL: NCT01383018
Title: Prospective Registry of Outcomes With Penile Prosthesis for Erectile Restoration (PROPPER)
Brief Title: PROPPER Prospective Registry of Outcomes With Penile Prosthesis
Acronym: PROPPER
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: U0552
Record Dates: First submitted 2011-06-24; First posted 2011-06-28 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction; Impotence
Keywords: Erectile Dysfunction (ED); Penile Implant; Impotence; Penile Prosthesis; Registry
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- AMS penile prosthesis receipients: Men for whom an AMS penile prosthesis is recommended
  Interventions: Device: AMS Penile Prosthesis Devices

INTERVENTIONS:
Device: AMS Penile Prosthesis Devices — Non-interventional device registry. Outcomes for patients receiving marketed AMS penile prosthesis devices.
  Other Names: AMS 700; AMS Ambicor; AMS Spectra

SUMMARY:
The purpose of this observational registry is to collect and better understand "real-world" outcomes for men undergoing penile implant surgery to treat erectile dysfunction.

DETAILED DESCRIPTION:
A prospective, multi-center, observational registry to be conducted at multiple sites throughout the United States and Canada, to collect "real-world" penile prosthetic outcomes according to investigators' standard of care. Using questionnaires as well as electronic data collection, investigating physicians will prospectively measure patient responses at regular intervals over a one- to five year period. The physician researchers have identified key metrics for the study including effectiveness, durability, complications, and patient satisfaction; quality of life will also be analyzed, being defined through several validated patient surveys.

ELIGIBILITY:
Inclusion Criteria:

Men diagnosed with erectile dysfunction (ED) for whom an AMS penile prosthesis is recommended by their physician are eligible for inclusion. Potentially eligible men should also meet the following inclusion criteria for study enrollment:

* Willing and able to provide written informed consent prior to enrollment (if applicable).
* Willing to be seen or contacted by phone by the investigator and answer at least 2 questions related to satisfaction and device use 1 year following implantation of an AMS penile prosthesis.

Exclusion Criteria:

- Men who are deemed by their physician to be not suitable for a penile implant will be excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with ED in the United States and Canada.
Sampling Method: Non-Probability Sample
Enrollment: 1457 (Actual)
Dates: Start 2011-06-13 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Henry, MD, Principal Investigator — Ark-LA-Tek; Anthony J. Bella, MD, Principal Investigator — University of Ottawa; Edward Karpman, MD, Principal Investigator — El Camino Urology Medical Group; LeRoy Jones, MD, Principal Investigator — Urology San Antonio Research PA; Bryan T Kansas, MD, Principal Investigator — The Urology Team; Brian Christine, MD, Principal Investigator — Urology Centers of Alabama; Kevin McVary, MD, Principal Investigator — SIU School of Medicine; James Hotaling, MD, Principal Investigator — University of Utah; Mohit Khera, MD, Principal Investigator — Baylor College of Medicine; Eugene Rhee, MD, Principal Investigator — Kaiser Permanente
Locations (11):
- United States (10):
  - Urology Centers of Alabama, Homewood, Alabama
  - El Camino Urology Medical Group, Mountain View, California
  - Kaiser Permanente, San Diego, California
  - SIU School of Medicine, Springfield, Illinois
  - Ark-LA-Tek, Bossier City, Louisiana
  - Lahey Clinic, Burlington, Massachusetts
  - The Urology Team, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - Urology San Antonio Research, PA, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
- University of Ottawa, Ottawa, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- AMS Penile Prosthesis Recipients: Men for whom an AMS penile prosthesis is recommended
  AMS Penile Prosthesis Devices: Non-interventional device registry. Outcomes for patients receiving marketed AMS penile prosthesis devices.
Period: Overall Study
Arm/Group | AMS Penile Prosthesis Recipients
Started | 1457
Completed | 1082
Not Completed | 375
Not completed — Adverse Event | 14
Not completed — Death | 10
Not completed — Lost to Follow-up | 5
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 9
Not completed — Subject not implanted | 76
Not completed — Missed Visit | 247
Not completed — Site closed early-not compliance related | 7
Not completed — Patient moved away from site | 1
Not completed — Subject Incarcerated | 1

BASELINE CHARACTERISTICS:
Population: AMS penile prosthesis recipients that completed baseline assessments. Subjects that started the study but did not have implantation are not included.
Arm/Group | AMS Penile Prosthesis Recipients
Number analyzed (Participants) | 1380
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1380
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77
  Not Hispanic or Latino | 1303
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 187
  White | 1152
  More than one race | 0
  Unknown or Not Reported | 20
Primary ED etiology [Count of Participants; unit: Participants]
  Radical prostatectomy (RP) | 369
  Diabetes | 283
  Cardiovascular disease | 251
  Peyronies disease | 123
  Priaprism | 19
  Other | 335

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Penile Prosthesis Overall Subject Satisfaction
Description: Penile prosthesis overall subject satisfaction (effectiveness objective 1) measured using a non-validated, standard question, evaluated overall and by penile prosthesis.
Time Frame: 1 year, post-implantation
Population: Subjects who received an AMS penile prosthesis and completed 1 year follow-up visit.
Measure: Count of Participants; unit: Participants
Groups:
- All AMS Penile Prosthesis Recipients - Total Reponses: Men for whom an AMS penile prosthesis is recommended
  AMS Penile Prostheses: Non-interventional device registry. Outcomes for subjects receiving a marketed AMS penile prosthesis.
- AMS 700: AMS 700, only
  Men for whom an AMS 700 penile prosthesis was recommended
- AMS Ambicor: AMS Ambicor, only
  Men for whom an AMS Ambicor penile prosthesis was recommended
- Spectra: Spectra, only
  Men for whom a Spectra penile prosthesis was recommended
Arm/Group | All AMS Penile Prosthesis Recipients - Total Reponses | AMS 700 | AMS Ambicor | Spectra
Number analyzed (Participants) | 1082 | 1050 | 21 | 11
Participants
  Very Dissatisfied | 34 | 34 | 0 | 0
  Dissatisfied | 37 | 35 | 2 | 0
  Neither Satisfied nor Dissatisfied | 71 | 68 | 2 | 1
  Satisfied | 297 | 286 | 5 | 6
  Very Satisfied | 643 | 627 | 12 | 4

2. Primary Outcome: Number of Participants With Penile Prosthesis That Are Using the Device
Description: Number of subjects using penile prosthesis at 1 year (effectiveness objective 1) measured using a non-validated, standard question, evaluated overall and by penile prosthesis.
Time Frame: 1 year, post implantation
Population: Subjects who received an AMS penile prosthesis and completed 1 year follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | All AMS Penile Prosthesis Recipients - Total Reponses | AMS 700 | AMS Ambicor | Spectra
Number analyzed (Participants) | 1082 | 1050 | 21 | 11
Participants | 984 | 956 | 18 | 10

3. Primary Outcome: Number of Participants With Penile Prosthesis That Are Using the Device Indicating How Often Their Use is.
Description: Penile prosthesis use at year (effectiveness objective 1) measured using a non-validated, standard question, evaluated overall and by penile prosthesis.
Time Frame: 1 year, post implantation
Population: Subjects who received an AMS penile prosthesis and completed 1 year follow-up visit who answered that they were using the device and responded to how often they were using it.
Measure: Count of Participants; unit: Participants
Arm/Group | All AMS Penile Prosthesis Recipients - Total Reponses | AMS 700 | AMS Ambicor | Spectra
Number analyzed (Participants) | 895 | 867 | 18 | 10
Participants
  Less than once per month | 58 | 56 | 1 | 1
  More than once per month | 837 | 811 | 17 | 9

4. Primary Outcome: Number of Times Per Month Participants With Penile Prosthesis Are Using the Device.
Description: Penile prosthesis use at 1 year measured in number of times per month (effectiveness objective 1) measured using a non-validated, standard question, evaluated overall and by penile prosthesis.
Time Frame: 1 year, post implantation
Population: Subjects who received an AMS penile prosthesis and completed 1 year follow-up visit who hand answered that they were using the device and responded to how many times per month they were using it.
Measure: Mean (Standard Deviation); unit: Number of times per month
Arm/Group | All AMS Penile Prosthesis Recipients - Total Reponses | AMS 700 | AMS Ambicor | Spectra
Number analyzed (Participants) | 490 | 467 | 17 | 6
Number of times per month | 6.3 (5.5) | 6.3 (5.6) | 5.4 (3.3) | 5.2 (4.3)

5. Primary Outcome: Number of Participants With Penile Prosthesis That Were Not Using the Device, Reasons for Non-use
Description: Penile prosthesis reasons for non-use at 1 year (effectiveness objective 1) measured using a non-validated, standard question, evaluated overall and by penile prosthesis.
Time Frame: 1 year, post implantation
Population: Subjects who received an AMS penile prosthesis and completed 1 year follow-up visit who had answered that they were not using the device and responded to the reason for non-use.
Measure: Count of Participants; unit: Participants
Arm/Group | All AMS Penile Prosthesis Recipients - Total Reponses | AMS 700 | AMS Ambicor | Spectra
Number analyzed (Participants) | 89 | 87 | 2 | 0
Participants
  Loss of partner | 8 | 7 | 1 | 0
  Partner disinterest | 9 | 8 | 1 | 0
  Device problem | 8 | 8 | 0 | 0
  Device dissatisfaction | 17 | 17 | 0 | 0
  Health decline | 13 | 13 | 0 | 0
  Other reason | 34 | 34 | 0 | 0

6. Primary Outcome: Number of Participants With Penile Prosthesis Using the Device But Not as Often as Desired
Description: Number of penile prosthesis subjects using the device but indicated that they were not using as often as desired (effectiveness objective 1) measured using a non-validated, standard question, evaluated overall and by penile prosthesis.
Time Frame: 1 year, post implantation
Population: Subjects who received an AMS penile prosthesis and completed 1 year follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | All AMS Penile Prosthesis Recipients - Total Reponses | AMS 700 | AMS Ambicor | Spectra
Number analyzed (Participants) | 1082 | 1050 | 21 | 11
Participants | 109 | 96 | 9 | 4

7. Primary Outcome: Number of Participants With Penile Prosthesis That Are Using the Device Less Than Desired or Dissatisfied - Reason Device Used Less Than Desired or Dissatisfied
Description: Reason why subject is using penile prosthesis less than desired or dissatisfied (effectiveness objective 1) measured using a non-validated, standard question, evaluated overall and by penile prosthesis.
Time Frame: 1 year, post implantation
Population: Subjects who received an AMS penile prosthesis and completed 1 year follow-up visit and responded that they were using the device less than desired or dissatisfied.
Measure: Count of Participants; unit: Participants
Arm/Group | All AMS Penile Prosthesis Recipients - Total Reponses | AMS 700 | AMS Ambicor | Spectra
Number analyzed (Participants) | 133 | 117 | 11 | 5
Participants
  Loss of partner | 4 | 4 | 0 | 0
  Partner disinterest | 9 | 8 | 0 | 1
  Device problem | 6 | 5 | 1 | 0
  Device dissatisfaction | 14 | 14 | 0 | 0
  Health decline | 13 | 12 | 1 | 0
  Other reason | 87 | 74 | 9 | 4

8. Other Pre Specified Outcome: Subject Reported 5-question International Index of Erectile Function (IIEF-5) Total Score, Baseline Through Five Years
Description: Penile prosthesis International Index of Erectile Function (IIEF-5) score (effectiveness objective 2) measured using a validated, multi-dimensional, self-administered questionnaire. Overall responses are reported. A higher score demonstrates an improvement in erectile function while a lower score indicates a loss of erectile function. The 5-question International Index of Erectile Function (IIEF-5) Questionnaire is a validated, multi-dimensional, self-administered investigation that has been found useful in the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials. A score of 0 to 5 is awarded to each of the 5 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire, and intercourse satisfaction. The subscales are summed to calculated the total score. The minimum total score for this questionnaire is 0 with a maximum of 30.
Time Frame: Baseline through 5 years
Population: Number of subjects analyzed reduced over time due to attrition. Also, follow-up after 1 year was optional.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All AMS Penile Prosthesis Recipients - Total Reponses: Men for whom an AMS penile prosthesis was recommended
  AMS Penile Prosthesis Devices: Non-interventional device registry. Outcomes for patients receiving a marketed AMS penile prosthesis.
Arm/Group | All AMS Penile Prosthesis Recipients - Total Reponses
Number analyzed (Participants) | 1194
score on a scale
  Baseline | 6.4 (5.2)
  1 year: number analyzed (Participants) | 853
  1 year | 20.6 (6.4)
  2 year: number analyzed (Participants) | 777
  2 year | 20.4 (6.6)
  3 year: number analyzed (Participants) | 595
  3 year | 21.2 (6.1)
  4 year: number analyzed (Participants) | 457
  4 year | 20.6 (6.8)
  5 year: number analyzed (Participants) | 291
  5 year | 21.2 (6.2)

9. Other Pre Specified Outcome: Erection Hardness Scale Over Five Years
Description: The Erection Hardness Scale (EHS), an easy-to-use, four-point scale for erectile dysfunction, provides a reliable measure of erection hardness and an indicator of other health and wellbeing outcomes, according to new data reported at the European Association of Urology. EHS rates the hardness of erection on a scale of zero to four, with four being the maximal score. A higher score indicates a harder penis while a lower score indicates greater dysfunction.
Time Frame: Baseline through 5 years
Population: Number of subjects analyzed reduced over time due to attrition. Also, follow-up after 1 year was optional.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All AMS Penile Prosthesis Recipients - Total Reponses
Number analyzed (Participants) | 1209
score on a scale
  Baseline | 1.0 (1.1)
  1 year: number analyzed (Participants) | 855
  1 year | 3.4 (1.0)
  2 year: number analyzed (Participants) | 779
  2 year | 3.5 (1.0)
  3 year: number analyzed (Participants) | 594
  3 year | 3.5 (0.9)
  4 year: number analyzed (Participants) | 462
  4 year | 3.5 (1.0)
  5 year: number analyzed (Participants) | 289
  5 year | 3.5 (0.9)

10. Other Pre Specified Outcome: American Urology Association - Symptom Index Over Five Years
Description: The AUA-SI contains seven symptoms questions which include feeling of incomplete bladder emptying, frequency, intermittency, urgency, weak stream, straining and nocturia, each referring to during the last month, and each involving assignment of a score from 0 to 5 for a total score of maximum 35 points from "non-missing" items. The lower score means a better quality of life.
Time Frame: Baseline through 5 years
Population: Number of subjects analyzed reduced over time due to attrition. Also, follow-up after 1 year was optional.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All AMS Penile Prosthesis Recipients - Total Reponses
Number analyzed (Participants) | 1114
score on a scale
  Baseline | 9.0 (6.9)
  1 year: number analyzed (Participants) | 805
  1 year | 7.9 (6.6)
  2 year: number analyzed (Participants) | 741
  2 year | 8.8 (7.0)
  3 year: number analyzed (Participants) | 564
  3 year | 8.2 (6.5)
  4 year: number analyzed (Participants) | 433
  4 year | 8.1 (6.3)
  5 year: number analyzed (Participants) | 281
  5 year | 8.1 (5.7)

11. Other Pre Specified Outcome: UCLA Prostate Cancer Index Over Five Years
Description: The University of California Los Angeles-Prostate Cancer Index -UCLA-PCI is a validated, twenty question questionnaire to asses impact of treatment for early stage prostate cancer on quality of life. The UCLA-PCI is analyzed in six sections, Sexual Function and Sexual Bother, Urinary Function and Urinary Bother, and Bowel Function and Bowel Bother. This is to measure not just the impact on function but also the quality of life impact. The UCLA PCI domain is scored on a scale of 0-100 points with higher values representing better outcomes.
Time Frame: Baseline through 5 years
Population: Number of subjects analyzed reduced over time due to attrition. Also, follow-up after 1 year was optional.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- UCLA-PCI Sexual Function: Sexual function measure
- UCLA-PCI Urinary Function: Urinary function measure
- UCLA-PCI Bowel Function: Bowel function measure
- UCLA-PCI Sexual Bother: Sexual bother measure
- UCLA-PCI Urinary Bother: Urinary bother measure
- UCLA-PCI Bowel Bother: Bowel bother measure
Arm/Group | UCLA-PCI Sexual Function | UCLA-PCI Urinary Function | UCLA-PCI Bowel Function | UCLA-PCI Sexual Bother | UCLA-PCI Urinary Bother | UCLA-PCI Bowel Bother
Number analyzed (Participants) | 833 | 814 | 804 | 820 | 812 | 802
score on a scale
  Baseline | 21.5 (16.9) | 79.9 (24.3) | 85.0 (15.5) | 10.8 (22.8) | 76.7 (31.6) | 85.5 (24.1)
  1 year: number analyzed (Participants) | 619 | 616 | 613 | 614 | 615 | 614
  1 year | 70.9 (20.9) | 82.6 (20.9) | 88.4 (14.3) | 77.3 (32.7) | 81.1 (26.6) | 87.3 (22.3)
  2 year: number analyzed (Participants) | 619 | 616 | 614 | 611 | 617 | 614
  2 year | 70.0 (21.6) | 83.4 (20.8) | 87.8 (15.9) | 77.9 (33.2) | 80.5 (27.3) | 86.5 (23.5)
  3 year: number analyzed (Participants) | 494 | 487 | 486 | 488 | 487 | 486
  3 year | 71.7 (20.8) | 83.8 (21.2) | 87.5 (17.1) | 78.8 (32.2) | 79.0 (28.3) | 86.8 (23.7)
  4 year: number analyzed (Participants) | 403 | 401 | 404 | 401 | 402 | 403
  4 year | 70.3 (22.2) | 86.0 (19.6) | 87.8 (17.3) | 80.7 (31.9) | 79.9 (27.3) | 86.6 (24.3)
  5 year: number analyzed (Participants) | 261 | 261 | 261 | 261 | 262 | 261
  5 year | 71.2 (21.3) | 85.9 (21.5) | 86.7 (19.3) | 83.1 (29.4) | 80.5 (28.3) | 84.8 (26.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all subjects who had the study device implanted through optional 5 year follow-up.
Description: All device and/or procedure related events were collected for this study.
Arm/Group | AMS Penile Prosthesis Receipients
All-Cause Mortality (participants affected / at risk) | 44/1380
Serious Adverse Events (participants affected / at risk) | 36/1380
Other Adverse Events (participants affected / at risk) | 72/1380
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMS Penile Prosthesis Receipients (N=1380)
Device Infection (Infections and infestations) | 11 (13) — 13 Device Infections, 10 were device related, 5 were procedure related, 3 of these were related to both device and procedure. All events were resolved.
Erosion (Injury, poisoning and procedural complications) | 6 (6) — 6 Erosion, 6 were device related with 2 being determined to also be procedure related All events were resolved.
Reservoir Herniation (Injury, poisoning and procedural complications) | 3 (3) — 3 Reservoir Herniation, 2 were device related, 1 was procedure related. All events were resolved.
Abscess (Infections and infestations) | 2 (2) — 2 Abscess, 2 were device related with 1 being determined to also be procedure related. All events were resolved.
Hematoma (Injury, poisoning and procedural complications) | 2 (2) — 2 Hematoma events, 2 were procedure related, 1 was related to both device and procedure.
Pain/Discomfort (Injury, poisoning and procedural complications) | 1 (1) — 1 Pain/Discomfort events, device related.
Urinary Retention (Renal and urinary disorders) | 2 (2) — 2 urinary retention events, 1 was procedure related and 1 was device related.
Cardiac Event - Non-specific (Vascular disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) — 1 cellulitis event, procedure related.
Cylinder Crossover (Injury, poisoning and procedural complications) | 1 (1) — 1 cylinder crossover event, device related
Device Cylinder Aneruysm/Bulge (Product Issues) | 1 (1) — 1 device cylinder aneurysm/bulge, device related
Edema - Scrotal (Skin and subcutaneous tissue disorders) | 1 (1) — 1 edema - scrotal event, procedure and device related.
Extrusion (Injury, poisoning and procedural complications) | 1 (1) — 1 extrusion event, device and procedure related
Pain/Discomfort - Penile (General disorders) | 1 (1) — 1 pain/discomfort-penile event, device and procedure related
Perforation - Other (Injury, poisoning and procedural complications) | 1 (1) — 1 perforation event, device related
Peyronie's Disease (Reproductive system and breast disorders) | 1 (1) — 1 Peyronie's Disease event, device related
Proximal Corporal Perforation (Injury, poisoning and procedural complications) | 1 (1) — 1 proximal corporal perforation event, procedure related
Pulmonary Embolus (Vascular disorders) | 1 (1) — 1 pulmonary embolus event, procedure event
Urethral Obstruction (Product Issues) | 1 (1) — 1 urethral obstruction event, device related
Would Dehiscence (Skin and subcutaneous tissue disorders) | 1 (1) — 1 wound dehiscence event, procedure related
Other - Substernal Chest Pain (Cardiac disorders) | 1 (1) — The event was reported by the site as not procedure or device related which does not fit the definition of a reportable SADE or UADE per the protocol.
Pain/Discomfort (General disorders) | 1 (1)
Other - Decreased Oxygen Saturation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMS Penile Prosthesis Receipients (N=1380)
Hematoma (Injury, poisoning and procedural complications) | 1 (1)
Urinary Retention (Injury, poisoning and procedural complications) | 3 (3)
Device Infection (Infections and infestations) | 5 (5)
Erosion (Injury, poisoning and procedural complications) | 5 (5)
Pain/Discomfort (General disorders) | 2 (2)
Reservoir Herniation (Injury, poisoning and procedural complications) | 4 (4)
Superficial Wound Infection (Infections and infestations) | 4 (4)
Device Cylinder Aneurysm/Bulge (Product Issues) | 3 (3)
Migration (pump) (General disorders) | 1 (1)
Urethral Trauma (Injury, poisoning and procedural complications) | 3 (3)
Extrusion (Injury, poisoning and procedural complications) | 2 (2)
Malposition (Product Issues) | 2 (2)
Pain/Discomfort - Groin (General disorders) | 1 (1)
Priapism (Reproductive system and breast disorders) | 1 (2)
Adhesion of the Pump/Scrotum (Skin and subcutaneous tissue disorders) | 1 (1)
Allergic reaction/Hypersensitivity Reaction (Immune system disorders) | 1 (1)
Auto Inflation (Product Issues) | 1 (1)
Bladder Neck Obstruction (Renal and urinary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Device Placement Failure (Injury, poisoning and procedural complications) | 1 (1)
Edema - Penile (Skin and subcutaneous tissue disorders) | 1 (1)
Fever (Investigations) | 1 (1)
Fibrosis (Product Issues) | 1 (1)
Fibrous Capsule Formation (Injury, poisoning and procedural complications) | 1 (1)
Hematospermia (Reproductive system and breast disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Incorrect Size - Cylinders too Large (Product Issues) | 1 (1)
Increased Blood Loss (Vascular disorders) | 1 (1)
Inguinal Hernia Formation (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain/Discomfort - Other (General disorders) | 1 (1)
Pain/Discomfort - Penile (General disorders) | 1 (1)
Pain/Discomfort With Erections (General disorders) | 1 (1)
Patient Dissatisfaction (General disorders) | 1 (1)
Perforation - Other (Injury, poisoning and procedural complications) | 1 (1)
Peyronie's Disease (Reproductive system and breast disorders) | 1 (1)
Proximal Corporal Perforation (Injury, poisoning and procedural complications) | 1 (1)
Urinary Tract Infection - UTI (Infections and infestations) | 1 (1)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 3 (3)
Pain/Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain/Discomfort (Product Issues) | 1 (1)
Migration (Pump) (Injury, poisoning and procedural complications) | 1 (1)
Migration (Pump) (Product Issues) | 1 (1)
Pain/Discomfort - Groin (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 2 (2)
Pain/Discomfort - Testicular (General disorders) | 1 (1)
Pain/Discomfort - Testicular (Product Issues) | 2 (2)
Other - Buckling of left cylinder led to left downward curvature (Product Issues) | 1 (1)
Other - Painful mass in right hemiscrotum (Reproductive system and breast disorders) | 1 (1)
Other - Left distal tip migration with pain at tip of penis with intercourse (Injury, poisoning and procedural complications) | 1 (1)
Other - Right cylinder protruding (Product Issues) | 1 (1)
Other - Pinching sensation around the resevoirs (General disorders) | 1 (1)
Other - Change in curvature of penis (increase in curvature) (Injury, poisoning and procedural complications) | 1 (1)
Other - Proximal cross over during IPP surgery (Injury, poisoning and procedural complications) | 1 (1)
Other - Incisional drainage (Infections and infestations) | 1 (1)
Other - Bilateral corporal aneurysm (Product Issues) | 1 (1)
Other - Proximal crossover (Injury, poisoning and procedural complications) | 1 (1)
Other - Slight separation of penoscrotal wound (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT01383018/Prot_SAP_000.pdf